CLINICAL TRIAL: NCT00181025
Title: Isolated Pelvic and Limb Perfusion With 1mg TNFa in the Treatment of Locally Advanced Sarcoma of Pelvis and Limbs' Girdle
Brief Title: Isolated Pelvic and Limb Perfusion in the Treatment of Locally Advanced Sarcoma of Pelvis and Limbs' Girdle
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIP; CSET 2003/1053
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2007-06-12 (Estimated); Status verified 2006-09

CONDITIONS: Sarcoma of Pelvis
Keywords: Limbs' girdle
MeSH Terms: interventions — Melphalan

INTERVENTIONS:
Drug: Tasonermine (TNFa)
Drug: Melphalan

SUMMARY:
This study looks at isolated pelvic perfusion and limbs' girdle with 1 mg tumor necrosis factor alpha (TNFa) in the treatment of locally advanced sarcoma of the pelvis and limbs' girdle.

ELIGIBILITY:
Inclusion Criteria:

* Soft tissue or bone sarcomas locally advanced of the pelvis or limbs' girdle

Exclusion Criteria:

* Resectable tumor without mutilation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2004-05

PRIMARY OUTCOMES:
Complete response rate on MRI

SECONDARY OUTCOMES:
Histological response
Objective responses
Rate of conservative treatments
Overall survival and disease free survival
Local and systemic toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Bonvalot, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave-Roussy, Villejuif, France